CLINICAL TRIAL: NCT04178135
Title: Recombinant LH Supplementation Timing Strategies (From Day 1 or Day 6) to a Standard GnRH Agonist Long Protocol in Subsequent COS Cycle of Older Patients With Unexpected Poor or Suboptimal Ovarian Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2019005
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility,Female
Keywords: poor or suboptimal ovarian response,GnRH agonist long protocol
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rLH supplementation from day 1 of stimulation (Experimental): rLH supplementation from day 1 of stimulation
  Interventions: Drug: rLH
- rLH supplementation from day 6 of stimulation (Active Comparator): rLH supplementation from day 6 of stimulation
  Interventions: Drug: rLH

INTERVENTIONS:
Drug: rLH — rLH supplement from day 1 of stimulation
  Arms: rLH supplementation from day 1 of stimulation
Drug: rLH — rLH supplement from day 6 of stimulation
  Arms: rLH supplementation from day 6 of stimulation

SUMMARY:
A randomized, controlled, pilot study, for Patients ≥ 35 years and < 40 years old with sufficient ovarian reserve parameters (AFC≥ 5), but showed an unexpected poor or suboptimal ovarian response(defined as ≤ 9 retrieved oocytes in previous full-stimulation cycle, but not get live birth after all embryos were used ). In order to get better oocyte number and quality in the new COS cycle, we will compare LH supplementation from beginning with from middle of stimulation in GnRH-a long protocol.

ELIGIBILITY:
Inclusion Criteria:

1.Infertile women, 35≤ Age< 40 years 2.18<BMI<28 Kg/m2 3.5 ≤AFC ≤20 4.Basal serum FSH≤10 IU/L, E2<70 pg/ml 5.Previous cycle as the first COS cycle,AFC ≥ 5,starting dose of FSH between 150 IU and 300IU with the possibility of adding r-hLH or hMG later in the cycle, number of oocytes retrieved ≤9 (4-9 oocytes retrieval as suboptimal responder and <4 oocytes retrieval as unexpected poor responder), but not get live birth after all embryos were used.

6.Normal uterus and at least one side of the normal ovary 7.GnRH-a long protocol, using Gonal-F® 300IU and Luveris® 150IU for COS 8.Informed consent form signed 9.Willing to follow the study protocol, and able to complete this study

Exclusion Criteria:

1. Moderate and Severe endometriosis
2. PCOS
3. Previous ovarian surgery history
4. History of recurrent miscarriages (>2 times of miscarriages)
5. Any major systemic disease that as per Investigator's discretion precludes subject for participation in the study
6. With pregnancy contraindications Alcoholism, drug abuse, drug addiction or patients with uncured sexually transmitted disease
7. According to the judgment of the Investigator, any medical condition or any concomitant surgery/medications that would interfere with evaluation of study medications
8. Simultaneous participation in another clinical study
9. Plan to use other Gn other than Gonal-F® or Luveris® during COS treatment Thyroid gland disorders

Ages: 35 Months to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of gestational sacs | Day 28 after embryo transfer
  Number of gestation sac will be detected by ultrasonographic visualization

CONTACTS AND LOCATIONS:
Overall Officials: Sufen Cai, Doctor, Principal Investigator — Reproductive and Genetic hospital of CITIC-xiangya
Locations (1):
- Reproductive & Genetic Hospital of CITIC-XIANGYA, Changsha, Hunan, China